CLINICAL TRIAL: NCT04058509
Title: Clinical Predictors of Extracorporal Shockwave Therapy Efficacy in Patients Presenting With Lateral Hip Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg University Hospital (Other)
Collaborators: University of Canberra (Other)
Responsible Party: Principal Investigator, Carsten Møller Poulsen Mølgaard, Clinical research physiotherapist, Aalborg University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N-20180036
Record Dates: First submitted 2019-08-14; First posted 2019-08-15 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Tendinopathy
Keywords: Greater Trochanter Pain Syndrome; Lateral hip pain
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- focused shockwave therapy (Experimental): 3 sessions of shock wave treatment.(Focused Shockwave Therapy).
  Interventions: Combination Product: Focused shockwave therapy

INTERVENTIONS:
Combination Product: Focused shockwave therapy — 3 session of shockwave therapy. The wave is focused through a standoff and transmitted into the tissue. Enhanced Energy: 0.01 - 0.55mJ/mm2. Broad Frequency Range: 1 - 8Hz. 12.5 cm penetration with pinpoint focus. The patient will be treated in the lateral decubitus position. The shock wave will focus on the area of maximal tenderness, which will be treated in a circumferential pattern.

SUMMARY:
This pragmatic clinical trial is considering the variable response to treatment outcome of individuals with Greater Trochanteric Pain Syndrome (GTPS). The aim of this study is to identify predictors of focused extracorporeal shockwave therapy (fESWT) efficacy in individuals with GTPS. Specifically, the ability of clinically applicable measurements including: Patient demographics, co-morbidity, oestrogen levels, pain characteristics, hip abductor strength, time to pain during single-leg stance test, low back pain, and immediate pain reduction to local anaesthetic injection at the trochanter major insertion of Gluteus medius (GMed) during walking.

ELIGIBILITY:
Inclusion Criteria:

* Lateral hip pain, worst over the greater trochanter, present for a minimum of 3 months
* Age 35-70 years
* Female
* Pain at an average intensity of ≥3 out of 10 on most days of the last week.
* Tenderness on palpation of the greater trochanter
* Pain on one of the following:

Reproduction of pain on 30 sec single leg stand OR Positive Faber test

Exclusion Criteria:

* Any known advanced hip joint pathology where groin pain is the primary complaint and/or reproduction of groin pain with Faber or FADDIR.
* Where range of pure hip joint flexion is <90°
* Radiating pain distal to the Gluteus Max + positive Straight Leg Raise (SLR-test < 30°)
* Known advanced knee pathology or restricted range of knee motion (must have minimum 90° flexion and full extension)
* Any systemic diseases affecting the muscular or nervous system, and uncontrolled diabetes
* Malignant tumour OR Systemic inflammatory disease
* Any factors that would preclude the participant from having an MRI (e.g. pacemaker, metal implants, pregnancy, claustrophobia)
* If the participant is involved in a legal/workcover or other injury claim
* Fear of needles (trypanophobia)
* If the participant is unable to write, read or comprehend Danish

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-11-28 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Global Rating of Change Scale | 3 months follow-up

SECONDARY OUTCOMES:
EuroQoL | 0, 12 and 26 weeks follow-up
  EQ-5D™
Muscle strength Static | 0, 12 and 26 weeks follow-up
  Hip abduction strength
Pain Pressure Threshold | 0, 12 and 26 weeks follow-up
  Lateral hip region
Patient-Specific Functional Scale). | 0, 6, 12 and 26 weeks follow-up
  difficulties with 1-5 functional tasks
PHQ9 | 0, 12 and 26 weeks follow-up
  Severity of depression
VISA-G | 0, 12 and 26 weeks follow-up
  disability score for gluteal tendinopathy

CONTACTS AND LOCATIONS:
Overall Officials: Carsten M Molgaard, PhD, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark